CLINICAL TRIAL: NCT04702529
Title: Soliton's Rapid Acoustic Pulse (RAP) Device for the Treatment of Fibrotic Scars: Multi-Treatment Proof-of-Concept Study
Brief Title: Treatment of Fibrotic Scars With Rapid Acoustic Pulse (RAP) Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soliton (Industry)
Collaborators: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-01
Record Dates: First submitted 2021-01-04; First posted 2021-01-11 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2023-05

CONDITIONS: Scars, Hypertrophic
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Three treatments to hypertrophic scar with RAP device (Experimental): RAP treatments will be administered to the scar every +/- 2 weeks for a total of 3 treatments
  Interventions: Device: Treatment of hypertrophic scars (Soliton's Rapid Acoustic Pulse (RAP) Device)

INTERVENTIONS:
Device: Treatment of hypertrophic scars (Soliton's Rapid Acoustic Pulse (RAP) Device) — Administration of 3 Rapid Acoustic Pulse (RAP) treatments

SUMMARY:
A multi-treatment proof of concept clinical study is to evaluate the safety, and efficacy of multiple treatments with Soliton's Rapid Acoustic Pulse (RAP) device for the improvement in the appearance of fibrotic scars

DETAILED DESCRIPTION:
Soliton's Rapid Acoustic Pulse(RAP) device is an electrohydraulic (EH) device using Soliton's Rapid Acoustic Pulse (RAP) technology developed to minimize the appearance of scars through both micro-disruption of the scar matrix leading to scar remodeling and down regulation of the 'fibrotic fibroblasts'

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years of age or older at the screening visit.
2. The participant is healthy, as determined by the investigator based on a medical evaluation including medical history.
3. The participant has a fibrotic scar (keloid or hypertrophic scar) that is easily delineated photographically located on the chest, back, trunk, upper arms or upper legs.
4. Scar must be located an essentially planar surface.
5. Scar size preferably between 2.5 cm2 and 5 cm2.
6. Preferably, the scar length is greater than 25 mm; and height greater than 2.5 mm.
7. Scar less than 5 years old.
8. Participant is willing to forego any other scar treatments until complete with study participation.
9. Participant is willing to participate in study and adhere to follow-up schedule.
10. Participant is able to read and comprehend English.

Regardless of the above, the final decision on scar inclusion will rest with the PI.

Exclusion Criteria:

1. Participant is sensitive to loud sounds
2. Participant had treatments, including topical steroids, to the scar being treated in the study in the prior 12 months.
3. Participant is unwilling to have research photos taken of treatment areas in the presence of Sponsor's researchers.
4. Participant is unwilling to have RAP treatment provided in the presence of Sponsor's researchers.
5. Participant is pregnant or planning to become pregnant during the duration of the study.
6. Metal or plastic implants near the area of the treatment (vascular stent, plates and screws, chest wires, hips, knees, elbows, etc.).
7. Active electronic implants such as pacemakers, defibrillators, cochlear implants, nerve/brain stimulators, drug pump, etc.
8. Medical disorder that would hinder the wound healing or immune response (no blood disorder, etc.).
9. History of coagulopathy(ies) and/or on anticoagulant medication.
10. Skin disorders (skin infections or rashes, extensive scarring, psoriasis, etc.) in the treatment area.
11. Current smoker.
12. Any surgical procedure in the prior 3 months, or planned during the duration of the study.
13. Any issue that, at the discretion of the Investigator, would interfere with assessment of safety or efficacy or compromise the participant's ability to fulfill study obligations
14. Treatment with another investigational device or agent within 30 days before treatment or during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Serious Adverse Events (SAEs) and Unexpected Adverse Events (UAEs) | Immediately post treatment
  Incidence of unexpected adverse events and serious adverse events directly attributable to the RAP device or treatment will be reported
Incidence of Treatment Emergent Serious Adverse Events (SAEs) and Unexpected Adverse Events (UAEs)Procedure Safety | up to 14 days
  Incidence of unexpected adverse events and serious adverse events directly attributable to the RAP device or treatment will be reported
Incidence of Treatment Emergent Serious Adverse Events (SAEs) and Unexpected Adverse Events (UAEs) | up to 3 week post treatment
  Incidence of unexpected adverse events and serious adverse events directly attributable to the RAP device or treatment will be evaluated before each treatment which occurs every 2 weeks, (+/- 1 week) and will be reported
Change from baseline scar Global Aesthetic Improvement Scale at 12 weeks | 12 weeks
  Noted improvement in scar appearance via Global Aesthetic Improvement Scale
  Scale (GAIS) as reported by the Principal Investigator (PI). Minimum value 1 and maximum value 5, with higher score meaning worse outcome.

SECONDARY OUTCOMES:
Change in baseline scar Global Aesthetic Improvement scale at 12 weeks | 12 weeks
  Noted improvement in scar via Patient and Observer Scar Assessment Scale (POSAS). Minimum value 1 and maximum value 10, with higher scores meaning a better outcome.
Change in baseline scar Global Aesthetic Improvement Scale at 12 weeks | 12 weeks
  Noted improvement in scar appearance via Global Aesthetic Improvement Scale (GAIS) as reported by the participant. Minimum value 1 and maximum value 5, with higher score meaning worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego Naval Medical Center, San Diego, California, United States